CLINICAL TRIAL: NCT06022224
Title: A Phase 2/3, Placebo-Controlled, Randomized, Observer-Blind Study To Evaluate the Safety, Tolerability, Immunogenicity, and Efficacy of a 2nd Generation E1/E2B/E3-Deleted Adenoviral COVID-19 Vaccine: The TCELL VACCINE TRIAL
Brief Title: A 2nd Generation E1/E2B/E3-Deleted Adenoviral COVID-19 Vaccine: The TCELL VACCINE TRIAL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: There were no participants enrolled into Phase 3 portion of the study because the study was prematurely terminated.
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID-3.001
Record Dates: First submitted 2023-08-30; First posted 2023-09-01 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The first 200 subjects randomized will comprise the phase 2 portion of the study.
  Enrollment may continue during this period and these subjects would be included in the phase 3 portion of the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- hAd5-S-Fusion+N-ETSD (Experimental): Prime (SC, Day 1) + Boost (SC, Day 22) @ 1x10^11 VP/dose
  Interventions: Biological: hAd5-S-Fusion+N-ETSD
- Placebo (Placebo Comparator): Prime (SC, Day 1) + Boost (SC, Day 22)
  Interventions: Biological: Placebo (0.9% (w/v) saline)

INTERVENTIONS:
Biological: hAd5-S-Fusion+N-ETSD — Clear and colorless liquid. Each vaccine is supplied in a 2-mL vial containing 1.0 mL of extractable vaccine at a concentration of 1 × 10^11 viral particles/mL.
  Arms: hAd5-S-Fusion+N-ETSD
Biological: Placebo (0.9% (w/v) saline) — Clear and colorless liquid.
  Arms: Placebo

SUMMARY:
This is a phase 2/3, multicenter, randomized, placebo-controlled, observer-blind study assessing the safety, tolerability, immunogenicity, and efficacy of prophylactic hAd5-S-Fusion+N-ETSD against COVID-19. It is intended that a minimum of 25% of subjects will be in the >55-year stratum. Safety, immunogenicity, and efficacy assessments will be conducted per the Schedule of Events (SoE) and subjects are expected to participate for up to a maximum of approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Male or female participants ≥16 years of age, at randomization.

   • Refer to Appendix 2 for reproductive criteria for male and female participants.

   Type of Participant and Disease Characteristics:
2. Participants who are willing and able to comply with all scheduled assessments, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

   Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included. Specific criteria for Phase 3 participants with known stable infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) can be found in Appendix 3.
4. Participants who, in the judgment of the investigator, are at higher risk for SARS-CoV-2 infection and subsequent development of COVID-19 (including, but not limited to, use of mass transportation, relevant demographics, and frontline essential workers).

   Informed Consent:
5. Capable of giving personal signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions:

1. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. Phase 2 only: Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
3. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
4. Receipt of medications intended to prevent COVID-19.
5. Previous clinical or microbiological diagnosis of COVID-19.
6. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
7. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate subcutaneous injection.
8. Women who are pregnant or breastfeeding.

   Prior/Concomitant Therapy:
9. Previous vaccination with any coronavirus vaccine.
10. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
11. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.

    Prior/Concurrent Clinical Study Experience:
12. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation. Other Exclusions
13. Investigator site staff or Sponsor employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 2 portion of the study enrolled participants. There were no participants enrolled into Phase 3 portion of the study because the study was prematurely terminated.
Groups:
- Phase 2 hAd5-S-Fusion+N-ETSD: Prime (SC, Day 1) + Boost (SC, Day 22) @ 1x10^11 VP/dose
  hAd5-S-Fusion+N-ETSD: Clear and colorless liquid. Each vaccine is supplied in a 2-mL vial containing 1.0 mL of extractable vaccine at a concentration of 1 × 10^11 viral particles/mL.
- Phase 2 Placebo: Prime (SC, Day 1) + Boost (SC, Day 22)
  Placebo (0.9% (w/v) saline): Clear and colorless liquid.
Period: Overall Study
Arm/Group | Phase 2 hAd5-S-Fusion+N-ETSD | Phase 2 Placebo
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hAd5-S-Fusion+N-ETSD | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (8.43) | 51.0 (18.12) | 53.1 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Healthy volunteers with no prior history of Covid [Count of Participants; unit: Participants] | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: To define the safety profile of prophylactic hAd5-SFusion+N-ETSD in the first 200 subjects randomized (Phase 2)
Time Frame: Up to 7 months (From day 1 to 6 months after last dose)
Population: Analysis population is all randomized subjects who received at least one dose of study intervention (safety analysis population)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 hAd5-S-Fusion+N-ETSD | Phase 2 Placebo
Number analyzed (Participants) | 17 | 18
Participants | 17 | 18

ADVERSE EVENTS:
Time Frame: From the time of first dose of study treatment until 1 month after the last dose of study treatment (including Assessment 3), up to 2 months. All SAEs were planned to be recorded by the investigator from the time of first dose of study treatment until 6 months after the last dose of study treatment, up to 7 months.
Groups:
- Prime (SC, Day 1) + Boost (SC, Day 22) @ 1x10^11 VP/Dose: hAd5-S-Fusion+N-ETSD
  : Clear and colorless liquid. Each vaccine is supplied in a 2-mL vial containing 1.0 mL of extractable vaccine at a concentration of 1 × 10^11 viral particles/mL.
- Prime (SC, Day 1) + Boost (SC, Day 22) Placebo (0.9% (w/v) Saline): Clear and Colorless Liquid: Placebo
- Group 1: hAd5-S-Fusion+N-ETSD; Group 1: Placebo: Solicited local reactogenicity adverse events from Day 1 through Day 7 after each vaccination
- Group 2: hAd5-S-Fusion+N-ETSD; Group 2:Placebo: Solicited systemic reactogenicity adverse events from Day 1 through Day 7 after each vaccination
- Group 3: hAd5-S-Fusion+N-ETSD; Group 3: Placebo: Unsolicited Adverse Events from First Vaccination through 7 Days after Last Vaccination
- Group 4: hAd5-S-Fusion+N-ETSD; Group 4: Placebo: Unsolicited Treatment Related Adverse Events First Vaccination through 7 Days after Last Vaccination
- Group 5: hAd5-S-Fusion+N-ETSD; Group 5: Placebo: Unsolicited Adverse Events from First Vaccination through 1 Month after Last Vaccination
- Group 6: hAd5-S-Fusion+N-ETSD; Group 6: Placebo: Unsolicited Treatment-Related Adverse Events First Vaccination through1 Month after Last Vaccination
- Group 7: hAd5-S-Fusion+N-ETSD; Group 7: Placebo: Serious Adverse Events from first Vaccination through 6 months after last Vaccination
Arm/Group | Prime (SC, Day 1) + Boost (SC, Day 22) @ 1x10^11 VP/Dose | Prime (SC, Day 1) + Boost (SC, Day 22) Placebo (0.9% (w/v) Saline): Clear and Colorless Liquid | Group 1: hAd5-S-Fusion+N-ETSD | Group 1: Placebo | Group 2: hAd5-S-Fusion+N-ETSD | Group 2:Placebo | Group 3: hAd5-S-Fusion+N-ETSD | Group 3: Placebo | Group 4: hAd5-S-Fusion+N-ETSD | Group 4: Placebo | Group 5: hAd5-S-Fusion+N-ETSD | Group 5: Placebo | Group 6: hAd5-S-Fusion+N-ETSD | Group 6: Placebo | Group 7: hAd5-S-Fusion+N-ETSD | Group 7: Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 17/17 | 5/18 | 12/17 | 7/18 | 15/17 | 3/18 | 15/17 | 1/18 | 15/17 | 3/18 | 15/17 | 1/18 | 0/17 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prime (SC, Day 1) + Boost (SC, Day 22) @ 1x10^11 VP/Dose (N=17) | Prime (SC, Day 1) + Boost (SC, Day 22) Placebo (0.9% (w/v) Saline): Clear and Colorless Liquid (N=18) | Group 1: hAd5-S-Fusion+N-ETSD (N=17) | Group 1: Placebo (N=18) | Group 2: hAd5-S-Fusion+N-ETSD (N=17) | Group 2:Placebo (N=18) | Group 3: hAd5-S-Fusion+N-ETSD (N=17) | Group 3: Placebo (N=18) | Group 4: hAd5-S-Fusion+N-ETSD (N=17) | Group 4: Placebo (N=18) | Group 5: hAd5-S-Fusion+N-ETSD (N=17) | Group 5: Placebo (N=18) | Group 6: hAd5-S-Fusion+N-ETSD (N=17) | Group 6: Placebo (N=18) | Group 7: hAd5-S-Fusion+N-ETSD (N=17) | Group 7: Placebo (N=18)
Injection site erythema (General disorders) | 0 | 0 | 15 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 16 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 12 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 9 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 7 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 15 | 0 | 15 | 0 | 15 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 11 | 0 | 11 | 0 | 11 | 0 | 0 | 0
Injection site warmth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 7 | 1 | 7 | 1 | 7 | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
There is an insufficient number of subjects enrolled to evaluate the efficacy of the Investigational Product. Thus, only safety results are provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT06022224/Prot_SAP_000.pdf